CLINICAL TRIAL: NCT00528307
Title: Changes in Myocardial Perfusion During Chronic Multi Site Biventricular Versus Right Ventricular Apex Pacing in Patients With Normal Left Ventricular Function Undergoing His Bundle Ablation for Drug-refractory Atrial Fibrillation
Acronym: SOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: R&D Cardiologie (Other)
Responsible Party: Principal Investigator, Vincent van Dijk, MD, R&D Cardiologie
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RDC-2006-03
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Atrial Fibrillation
Keywords: myocardial perfusion; His ablation; biventricular pacing; His bundle ablation for atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): First 3 months of biventricular pacing, second 3 months right ventricular apical pacing
  Interventions: Device: HIS buldle ablation
- 2 (Active Comparator): First 3 months of right ventricular apical pacing, second 3 months biventricular pacing
  Interventions: Device: HIS buldle ablation

INTERVENTIONS:
Device: HIS buldle ablation — HIS bundle ablation, followed by implant of a biventricular pacemaker

SUMMARY:
To determine whether Biventricular pacing in patients undergoing HIS bundle ablation for atrial fibrilation has beneficial effects on myocardial perfusion and left ventricularr ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Normal to nearly normal LVF (EF > 40%)
* Drug-refractory, persistent or permanent atrial fibrillation
* Referred for His ablation

Exclusion Criteria:

* Unwilling or unable to sign the informed consent
* Life expectancy < 1year from non-cardiac causes
* Previous myocardial infarction
* Previous coronary bypass surgery
* Poor left ventricle function (EF< 40%) from any cause
* Symptomatic obstructive coronary artery disease
* Poor ultra sound imaging quality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Difference in size of myocardial perfusion abnormalities in the two treatment groups as measured with MPS. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lucas VA Boersma, MD, PHD, Principal Investigator — St. Antonius Hospital
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands